CLINICAL TRIAL: NCT07216443
Title: A Phase 2 Trial of Orca-T Following Reduced Intensity or Nonmyeloablative Conditioning in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Trial of Orca-T Following Reduced Intensity or Nonmyeloablative Conditioning in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SERENE-T
Record Dates: First submitted 2025-09-29; First posted 2025-10-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Mixed Phenotype Acute Leukemia
Keywords: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Mixed Phenotype Acute Leukemia; Therapy-Related Myelodysplastic Syndrome; Hematopoietic Stem Cell Transplantation; Humans; Graft vs Host Disease; SERENE-T; ORCA-T; Disease; Pathologic Processes; Neoplasms by Histologic Type; Neoplasms; Hematologic Diseases; Bone Marrow Diseases; Precancerous Conditions; Neoplasms by Site; Disease Attributes; Immunoproliferative Disorders; Immune System Diseases; Leukemia; Preleukemia; Hematologic Neoplasms; Syndrome; Acute Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Biphenotypic, Acute; Graft vs Host Disease; Disease; Pathologic Processes; Neoplasms by Histologic Type; Neoplasms; Hematologic Diseases; Bone Marrow Diseases; Precancerous Conditions; Neoplasms by Site; Disease Attributes; Immunoproliferative Disorders; Immune System Diseases; Leukemia; Preleukemia; Hematologic Neoplasms; Syndrome; Acute Disease

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label phase 2 trial of Orca-T in adults with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) who are eligible for RIC-alloHCT or NMA-alloHCT with an 8/8 HLA-matched related or unrelated donor. Participants will receive Orca-T after the investigator's choice from the RIC and NMA regimens allowed as per protocol. Single-agent GVHD prophylaxis with tacrolimus will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orca-T (Experimental): Participants will receive [RIC or NMA conditioning] + Orca-T + single-agent tacrolimus based on eligibility and investigator's choice of conditioning regimen.
  Interventions: Biological: Orca-T

INTERVENTIONS:
Biological: Orca-T — An allogeneic stem cell and T-cell immunotherapy biologic

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of Orca-T in participants undergoing reduced intensity or non-myeloablative allogeneic hematopoietic cell transplantation (alloHCT) for hematologic malignancies. Orca-T is an allogeneic stem cell and T-cell immunotherapy biologic manufactured for each patient (transplant recipient) from the mobilized peripheral blood of a specific, unique donor. It is composed of purified hematopoietic stem and progenitor cells (HSPCs), purified regulatory T cells (Tregs), and conventional T cells (Tcons).

DETAILED DESCRIPTION:
This study is a multicenter, open-label phase 2 trial of Orca-T in adults with acute myeloid leukemia or myelodysplastic syndrome who are not able to receive myeloablative (high intensity) conditioning and are eligible for reduced intensity conditioning (RIC)-alloHCT or non-myeloablative (NMA)-alloHCT with an 8/8 human leukocyte antigen (HLA)-matched related or unrelated donor. The trial is designed to further characterize the safety and tolerability of Orca-T and to perform an initial assessment of the efficacy of Orca-T in participants eligible for RIC-alloHCT or NMA-alloHCT.

Participants will receive Orca-T after the investigator's choice from the RIC and NMA regimens followed by single-agent graft-versus-host disease (GVHD) prophylaxis with tacrolimus.

Prior to the initiation of this study (the SERENE-T Study), a phase 1 study (clinicaltrials.gov number: NCT05088356) was conducted to examine the safety and efficacy of Orca-T in participants receiving RIC-alloHCT. Participants have also been treated previously with Orca-T during an ongoing phase 1b/3 study (NCT05316701 and NCT04013685) in participants receiving a MAC regimen. The results of these studies have prompted Orca Bio to further evaluate Orca-T in participants receiving RIC or NMA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of enrollment
2. Diagnosed with 1 of the following diseases:

   1. Acute myeloid, or mixed phenotype leukemia in complete remission (CR) or CR with incomplete hematologic recovery (CRi), with or without the presence of known minimal residual disease.
   2. Myelodysplastic syndrome that is indicated for alloHCT per the 2017 International Expert Panel recommendations and/or therapy-related/secondary MDS as defined by the World Health Organization (WHO) classification of myeloid malignancies, with ≤10% blast burden in the bone marrow.
3. Planned to undergo 1 of the following preparative regimens as per Investigator discretion:

   1. RIC cohort: Planned RIC-alloHCT including RIC regimen with TBI/thiotepa/fludarabine
   2. NMA cohort: Planned NMA-alloHCT including NMA regimen with fludarabine/cyclophosphamide/TBI
4. Identified related or unrelated donor who is an 8/8 match for HLA-A, -B, -C, and -DRB1
5. Estimated glomerular filtration rate ≥30 mL/minute
6. Cardiac ejection fraction at rest ≥40% or shortening fraction of ≥22% by echocardiogram or radionuclide scan (MUGA)
7. Diffusing capacity of the lung for carbon monoxide (adjusted for hemoglobin) ≥40%
8. Negative serum or urine β-HCG test in persons of childbearing potential
9. Alanine transaminase (ALT)/aspartate transaminase (AST) <5 times the upper limit of normal (ULN)
10. Total bilirubin <3 × ULN
11. Deemed ineligible for a fully myeloablative alloHCT per assessment of the principal investigator

Exclusion Criteria:

1. Prior alloHCT
2. Currently receiving corticosteroids or other immunosuppressive therapy. Topical corticosteroids or oral systemic corticosteroid doses less than or equal to 10 mg/day are allowed.
3. Planned donor lymphocyte infusion (DLI)
4. Planned pharmaceutical in vivo or ex vivo T-cell depletion
5. Recipient-positive antidonor HLA antibodies against a mismatched allele in the selected donor
6. Karnofsky performance score <60%
7. For RIC cohort only: HCT-Specific Comorbidity Index (HCT-CI) ≥6
8. Uncontrolled bacterial, viral, or fungal infection (currently taking antimicrobial therapy and with progression or no clinical improvement) at the time of enrollment
9. Seropositive for HIV-1 or -2, HTLV-1 or -2, hepatitis B surface antigen, or HCV antibody unless previously treated with curative therapy and are HCV NAT negative
10. Known allergy or hypersensitivity to or intolerance of tacrolimus
11. Documented allergy or hypersensitivity to iron dextran or bovine, murine, algal, or Streptomyces avidinii proteins
12. Any uncontrolled autoimmune disease requiring active immunosuppressive treatment
13. Concurrent malignancy within 1 year except nonmelanoma skin cancer that has been curatively resected
14. Psychosocial circumstances that preclude the participant being able to go through transplantation or participate responsibly in follow-up care
15. Persons who are pregnant or breastfeeding
16. Person of childbearing potential (POCBP) or men who have sexual contact with POCBP who are unwilling to use effective forms of birth control or abstinence for 1 year after transplantation.
17. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's or medical monitor's judgment, precludes the recipient's safe participation in and completion of the trial or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
RIC Cohort: GVHD-free and relapse-free survival (GRFS) | Day 0 through day +365 after transplantation
  GRFS is defined as the time from the date of transplantation to the date of death from any cause, relapse, the first onset of grade 3 or 4 acute GVHD (graded per MAGIC criteria), or the first onset of moderate or severe chronic GVHD (graded per NIH consensus criteria), whichever is earliest.
NMA Cohort: Incidence of neutrophil engraftment | Day 0 through day +28 after transplantation
  Incidence of neutrophil engraftment is defined as achieving an ANC ≥500/mm3 for 3 consecutive days by day +28. The first of the 3 days will be designated the day of engraftment. If the ANC never drops below 500/mm3, day +1 will be designated the day of engraftment.
NMA Cohort: Time to neutrophil engraftment | Day 0 through day +28 after transplantation
  The first of the 3 days will be designated the day of engraftment. If the ANC never drops below 500/mm3, day +1 will be designated the day of engraftment.

SECONDARY OUTCOMES:
Safety of Orca-T | Day 0 through day +100 after transplantation
  The incidence of graft failure, grade ≥3 acute GVHD (per MAGIC criteria), grade ≥4 infection (per CTCAE v5.0), manufacturing failure, and non-relapse mortality for each cohort.
Incidence of serious infections | Day 0 through day +365 after transplantation
  The incidence of grade ≥3 infection (per CTCAE v5.0)
Severity of serious infection | Day 0 through day +365 after transplantation
  The severity of grade ≥3 infection (per CTCAE v5.0)
Overall survival | Day 0 through day +730 after transplantation
  The rate of overall survival for each cohort.
Non-relapse mortality | Day 0 through day +730 after transplantation
  The rate of non-relapse mortality for each cohort
Relapse-free survival | Day 0 through day +730 after transplantation
  The rate of relapse-free survival for each cohort.
Chronic GVHD-free survival | Day 0 through day +730 after transplantation
  The rate of chronic GVHD-free survival for each cohort
GVHD-free and relapse-free survival (GRFS) | Day 0 through day +730 after transplantation
  The rate of GRFS for the NMA cohort.
Incidence of acute GVHD | Day 0 through day +180 after transplantation
  The incidence of acute GVHD (all grades) for each cohort
Severity of acute GVHD | Day 0 through day +180 after transplantation
  The severity of acute GVHD (all grades) for each cohort
Time to onset of acute GVHD | Day 0 through day +180 after transplantation
  Time to first onset of grade 2 through 4 acute GVHD
Incidence of chronic GVHD | Day 0 through day +730 after transplantation
  The incidence of chronic GVHD (all grades)
Severity of chronic GVHD | Day 0 through day +730 after transplantation
  The severity of chronic GVHD (all grades)
Time to onset of acute GVHD | Day 0 through day +730 after transplantation
  Time to first onset of moderate or severe chronic GVHD
RIC cohort: Incidence of neutrophil engraftment | Day 0 through day +28 after transplantation
  The incidence of neutrophil engraftment in the RIC cohort.
RIC cohort: Time to neutrophil engraftment | Day 0 through day +28 after transplantation
  Time to neutrophil engraftment in the RIC cohort.
Incidence of platelet engraftment | Day 0 through day +50 after transplantation
  The incidence of platelet engraftment.
Time to platelet engraftment | Day 0 through day +50 after transplantation
  Time to platelet engraftment.
Incidence of steroid-refractory acute GVHD | Day 0 through day +180 after transplantation
  The incidence of steroid-refractory acute GVHD for each cohort.
Incidence of steroid-refractory chronic GVHD | Day 0 through day +730 post-transplant
  The incidence of steroid-refractory chronic GVHD for each cohort.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Department of Medicine, Los Angeles, California
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No